CLINICAL TRIAL: NCT03970681
Title: Clinical and Radiological Evaluation of Acoustic Neuromas With Spontaneous Shrinkage
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7417
Record Dates: First submitted 2019-05-29; First posted 2019-05-31 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Neuroma, Acoustic
Keywords: Acoustic neuroma; Vestibular schwannoma; Spontaneous shrinkage; Neoplasm regression; Volume quantification; Tridimensional measurements; Volumetric measurements
MeSH Terms: conditions — Neuroma, Acoustic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the regression characteristics of this Acoustic Neuroma population using volumetric data To study the relationship between regression and clinical characteristics including tinnitus, dizziness, hearing loss, and the intrinsic characteristics of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Major subject (≥18 years old)
* Subject followed in radiology for the assessment or follow-up of neuroma between January 01, 2013 and June 30, 2018
* Subject who has agreed to the use of his data for the purpose of this research
* Subject presenting an untreated neuroma

Exclusion Criteria:

* Subject having expressed his opposition to participating in the study
* Subject followed for neuroma of other cranial pairs,
* Subject followed in the context of type II neurofibromatosis
* Subject with a treated neuroma (radiotherapy or surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject followed in radiology for the assessment or follow-up of neuroma between January 01, 2013 and June 30, 2018
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-05-29 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Measurement of tumoral volume using tridimensional reconstruction on MRI, and kinetics of decay | Files analyzed from January 01, 2013 to June 30, 2018

CONTACTS AND LOCATIONS:
Locations (1):
- Service D'Orl Et de Chirurgie Cervico-Faciale, Strasbourg, France